CLINICAL TRIAL: NCT04540510
Title: Oscillatory Positive Expiratory Pressure Devices in Acute Inpatient Treatment of Pneumonia
Brief Title: OPEP Devices in Acute Inpatient Treatment of Pneumonia
Acronym: OPEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to COVID-19
Sponsor: Danbury Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-1104
Record Dates: First submitted 2020-08-28; First posted 2020-09-07 (Actual); Results first posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-08

CONDITIONS: Community-acquired Pneumonia
Keywords: Oscillatory positive expiratory pressure
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients randomized to the OPEP therapy added to standard pneumonia care OR standard pneumonia care..
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- OPEP therapy added to standard pneumonia care (Active Comparator): The intervention group will be asked to use an OPEP device twice daily, with the help of study investigators, for a total of at least 5 minutes per session. This treatment will be in addition to the usual care that the hospital physician prescribe for them to treat the pneumonia.
  Interventions: Device: OPEP therapy; Other: Standard care
- Standard pneumonia care (Active Comparator): The control group will continue to receive the usual care that their hospital team prescribe for them to treat the pneumonia.
  Interventions: Other: Standard care

INTERVENTIONS:
Device: OPEP therapy — Oscillatory Positive Expiratory Pressure therapy
  Arms: OPEP therapy added to standard pneumonia care
Other: Standard care — Standard pneumonia care

SUMMARY:
This is a randomized-controlled prospective study to be conducted at Danbury Hospital and Norwalk Hospital to evaluate oscillatory positive expiratory pressure (OPEP) devices for "airway clearance" (helping to clear out phlegm or mucous from your lungs and bronchial tubes) in the treatment of patients admitted to the hospital with pneumonia.

Approximately 200 subjects are expected to participate in this study.

DETAILED DESCRIPTION:
Pneumonia is one of the most common health conditions leading to hospitalization today. Approximately 1.3 million people in the US are admitted to the hospital with community-acquired pneumonia (CAP) annually, with readmission rates within the first 30 days as high as 20%. In a retrospective analysis of patients with culture-confirmed bacterial pneumonia, 30-day readmission occurred in 19.3% of patients. At Norwalk Hospital, the 30-day readmission rate for patients with pneumonia is 13.1%. CAP is the sixth most common cause of death with a case-fatality rate of up to 16% for hospitalized CAP patients, and an overall 30-day mortality up to 23%. The economic burden of CAP is also high, l with a CAP cost burden estimated to be at least $13 billion in 2008 within just the Medicare population.

There have been several small studies done to analyze the utility of airway clearance and its potential role in CAP. These studies have generally been small and have used a wide variety of airway clearance devices and techniques, including external chest wall physiotherapy devices and postural drainage, both now considered second line therapies for most patients. These studies have been variable in their findings and overall have not shown that airway clearance is either beneficial or harmful in CAP. The studies did show, however, that the duration of fever and hospital length of stay were both significantly decreased, suggesting the possibility of other clinically important benefits.

In this prospective randomized controlled trial, investigators will test the hypothesis that the use of OPEP devices, specifically the handheld Aerobika (Monaghan Medical) will result in more rapid and durable recovery in patients hospitalized with community-acquired pneumonia as measured by decreased hospital length of stay, reduced duration of fever, improvement in dyspnea, decreased duration of antibiotics, increased rate of diagnosis of the etiologic organism responsible for the pneumonia, and reduced readmission rates:

Primary outcome

1. Reduction in hospital length of stay

Secondary outcomes

1. Reduction in dyspnea by modified-Borg score
2. Reduction in duration of antibiotics
3. Reduction in duration of fever
4. Reduction in need for oxygen at hospital discharge
5. Reduction in 30-, 60-, and 90-day readmission rates
6. Diagnosis of organism by sputum
7. Transfer to the intensive care unit (ICU)

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms suggesting pneumonia (eg. cough, fever, pleuritic chest pain, sputum production, dyspnea)
* Any new chest radiographic infiltrate consistent with pneumonia

Exclusion Criteria:

* Untreated or recently (within the past 90 days) treated pneumothorax
* Active hemoptysis
* Recent facial, oral, or skull trauma
* Hemodynamically unstable patients
* Severe nausea or active vomiting
* Recent diagnosis of pneumonia prior to current inpatient encounter (within 60 days)
* Significant cognitive impairment or psychiatric conditions that prevent ability to participate in or cooperate with oPEP use
* Active TB or in negative pressure room
* Pregnancy
* Pre-existing medical condition with a life expectancy of less than 3 months
* Inability to form appropriate mouth seal on device (eg. due to neuromuscular disease)
* Pre-existing active use of oPEP devices
* Requiring >=50% FiO2 or facemask (excluding high flow NC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Ahasic, MD, Principal Investigator — Nuvance Health
Locations (1):
- Norwalk Hospital, Norwalk, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang M, Yan Y, Yin X, Wang BY, Wu T, Liu GJ, Dong BR. Chest physiotherapy for pneumonia in adults. Cochrane Database Syst Rev. 2013 Feb 28;(2):CD006338. doi: 10.1002/14651858.CD006338.pub3. PMID 23450568
- [Background] Narula D, Nangia V. Use of an oscillatory PEP device to enhance bronchial hygiene in a patient of post-H1NI pneumonia and acute respiratory distress syndrome with pneumothorax. BMJ Case Rep. 2014 Mar 7;2014:bcr2013202598. doi: 10.1136/bcr-2013-202598. PMID 24717858
- [Background] Graham WG, Bradley DA. Efficacy of chest physiotherapy and intermittent positive-pressure breathing in the resolution of pneumonia. N Engl J Med. 1978 Sep 21;299(12):624-7. doi: 10.1056/NEJM197809212991203. PMID 355879
- [Background] Christensen EF, Nedergaard T, Dahl R. Long-term treatment of chronic bronchitis with positive expiratory pressure mask and chest physiotherapy. Chest. 1990 Mar;97(3):645-50. doi: 10.1378/chest.97.3.645. PMID 2106412
- [Background] Halm EA, Fine MJ, Marrie TJ, Coley CM, Kapoor WN, Obrosky DS, Singer DE. Time to clinical stability in patients hospitalized with community-acquired pneumonia: implications for practice guidelines. JAMA. 1998 May 13;279(18):1452-7. doi: 10.1001/jama.279.18.1452. PMID 9600479
- [Background] Sato R, Gomez Rey G, Nelson S, Pinsky B. Community-acquired pneumonia episode costs by age and risk in commercially insured US adults aged >/=50 years. Appl Health Econ Health Policy. 2013 Jun;11(3):251-8. doi: 10.1007/s40258-013-0026-0. PMID 23605251
- [Background] File TM Jr, Marrie TJ. Burden of community-acquired pneumonia in North American adults. Postgrad Med. 2010 Mar;122(2):130-41. doi: 10.3810/pgm.2010.03.2130. PMID 20203464
- [Background] Khoudigian-Sinani S, Kowal S, Suggett JA, Coppolo DP. Cost-effectiveness of the Aerobika* oscillating positive expiratory pressure device in the management of COPD exacerbations. Int J Chron Obstruct Pulmon Dis. 2017 Oct 19;12:3065-3073. doi: 10.2147/COPD.S143334. eCollection 2017. PMID 29089755
- [Background] De Alba I, Amin A. Pneumonia readmissions: risk factors and implications. Ochsner J. 2014 Winter;14(4):649-54. PMID 25598730

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OPEP Therapy Added to Standard Pneumonia Care | Standard Pneumonia Care
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPEP Therapy Added to Standard Pneumonia Care | Standard Pneumonia Care | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (20.0) | 78.2 (11.3) | 77 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 37.4 (0.8) | 24.7 (3.0) | 30.4 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay
Description: Number of days that the patient stays in hospital was collected from medical record. We have calculated the mean and the standard deviation for both groups.
Time Frame: duration of hospital stay, an expected average of 4 days
Population: Although 6 subjects were recruited in the control group, however, we are missing this variable in data collection sheet for one subject in the control group. Therefore, we have only evaluated 5 subjects in the control group for this analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | OPEP Therapy Added to Standard Pneumonia Care | Standard Pneumonia Care
Number analyzed (Participants) | 5 | 5
days | 1.2 (0.9) | 4.0 (1.2)

2. Secondary Outcome: Reported Dyspnea by Modified-Borg Score
Description: Dyspnea as measured by modified-Borg score, minimum value 0 (No shortness of breath) and maximum value 10 (Maximal breathlessness). Score scale is from 0-10. We have calculated the mean and the standard deviation for both groups.
Time Frame: duration of hospital stay, an expected average of 4 days
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | OPEP Therapy Added to Standard Pneumonia Care | Standard Pneumonia Care
Number analyzed (Participants) | 5 | 6
score on scale | 1.2 (3.8) | 2.4 (2.0)

3. Secondary Outcome: Duration of Antibiotics
Description: Duration of antibiotics was collected from medical record. We have calculated the mean and the standard deviation for both groups.
Time Frame: duration of hospital stay, an expected average of 4 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | OPEP Therapy Added to Standard Pneumonia Care | Standard Pneumonia Care
Number analyzed (Participants) | 5 | 5
days | 8.8 (4.5) | 7.4 (4.3)

4. Secondary Outcome: Duration of Fever
Description: Duration of fever was collected from medical record. We have calculated the mean and the standard deviation for both groups.
Time Frame: duration of hospital stay, an expected average of 4 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | OPEP Therapy Added to Standard Pneumonia Care | Standard Pneumonia Care
Number analyzed (Participants) | 5 | 6
days | NA (NA) — no participants in the Treatment Group had fever | 0.8 (1.0)

5. Secondary Outcome: Number of Participants With Need for Oxygen Supplement at Hospital Discharge
Description: Number of participants with need for oxygen supplement at the time of hospital discharge was collected from medical record for both groups.
Time Frame: duration of hospital stay, an expected average of 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | OPEP Therapy Added to Standard Pneumonia Care | Standard Pneumonia Care
Number analyzed (Participants) | 5 | 6
Participants | 0 | 0

6. Secondary Outcome: Reported 30-, 60-, and 90-day Readmission Rates
Description: Number of total hospital readmissions post-enrollment was obtained from medical record.
Time Frame: 90 day after the hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | OPEP Therapy Added to Standard Pneumonia Care | Standard Pneumonia Care
Number analyzed (Participants) | 5 | 6
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Positive Sputum Culture
Description: Data on the diagnosis of organism by sputum (positive sputum culture) was collected from medical record. We have counted number of participants with intervention and without intervention.
Time Frame: duration of hospital stay, an expected average of 4 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | OPEP Therapy Added to Standard Pneumonia Care | Standard Pneumonia Care
Number analyzed (Participants) | 5 | 5
Participants | 1 | 3

8. Secondary Outcome: Number of Participants Transferred to the Intensive Care Unit (ICU)
Description: Number of participants transferred to the intensive care unit post enrollment was obtained from medical record for both groups.
Time Frame: duration of hospital stay, an expected average of 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | OPEP Therapy Added to Standard Pneumonia Care | Standard Pneumonia Care
Number analyzed (Participants) | 5 | 6
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each subject from the time informed consent was signed until termination from the study, up to a week
Arm/Group | OPEP Therapy Added to Standard Pneumonia Care | Standard Pneumonia Care
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT04540510/Prot_SAP_000.pdf